CLINICAL TRIAL: NCT00140517
Title: Relationships Between the Use of Antimalarial Drugs in Pregnancy and Plasmodium Falciparum Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: DBL -Institute for Health Research and Development (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HSR/DD/677-01/DG-CM/624-02
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria in Pregnancy; Birth Weight; Anaemia
Keywords: Plasmodium falciparum; malaria; pregnancy; resistance
MeSH Terms: conditions — Birth Weight; Anemia; Malaria, Falciparum; Malaria | interventions — fanasil, pyrimethamine drug combination; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: sulphadoxine-pyrimethamine
Drug: chloroquine

SUMMARY:
Plasmodium falciparum resistance to chloroquine (CQ) and sulfadoxine-pyrimethamine (SP) continue to spread, impeding control of this important disease. CQ and SP are still the most commonly used antimalarial drugs for malaria prevention during pregnancy and might be made less effective by resistance. However, the treatment and prophylaxis regimens used may also create conditions for selecting resistant malaria parasite strains. A better understanding of the relationships between chemoprophylaxis regimens and resistance would be helpful to improve chemoprophylaxis of malaria in pregnancy.

This work aims to improve the use of chemoprophylaxis in pregnancy by determining whether there is a relationship between the use of standard prophylactic regimens with CQ and SP and the occurrence of P. falciparum resistant strains in pregnant women. The study consists of 2 parts. The first part is a randomized trial comparing 3 chemoprophylactic treatment groups: - weekly CQ after initial presumptive CQ treatment, - CQ intermittent presumptive treatment given as a standard dose at 2nd and 3rd trimester, respectively and SP intermittent presumptive treatment given as a single dose at 2nd and 3rd trimester, respectively. These treatment groups will also be compared to a group of women delivering at the same health centre but who have not been participating in the study. The second part will be a clinical trial for assessment of clinical and parasitological efficacy of CQ and SP treatment in pregnant women presenting with uncomplicated malaria attacks.

The study will be conducted from October 2002 to March 2005 in a health centre of Ouagadougou, Burkina Faso where malaria transmission is seasonal and resistance to CQ and SP is low.

DETAILED DESCRIPTION:
OBJECTIVES Overall objective: To improve the use of malaria chemoprophylaxis in pregnancy.

Specific objectives:

To investigate the effects of weekly CQ, intermittent presumptive treatment with CQ, and with SP on placental, peripheral, and cord parasitaemia and on P. falciparum resistance status in primigravidae and secundigravidae.

To determine the relationships between carriage of P. falciparum resistant strains and malaria morbidity (attacks and anaemia) during pregnancy.

To determine the clinical and parasitological efficacy of CQ and SP in primigravidae and secundigravidae.

MATERIAL AND METHODS

The study will be conducted in a peripheral health centre of Ouagadougou, Burkina Faso, West Africa.

The largest part of the country is tropical savannah with a rainy season from June to October (average rainfall: 1000 mm per year, mean temperature > 25°C), a cold dry season from November to February, (min. temp. 15°C) and a hot dry season from March to May. Malaria transmission is seasonal (June to December)and the major mosquito vectors are A. gambiae, A. funestus and A. arabiensis. Malaria morbidity represents 30 to 50% of febrile illnesses and is the most frequent reason for health centres attendance and hospitals admission.Since it's first notification in 1986, P. falciparum resistance to CQ increased slowly with a considerable variation in space and time and resistance to SP has remained low. CQ clinical failures are in general less than 20% in 6-59 months children and parasitological resistance is around 30%. Malaria prevention in pregnancy is given as weekly 300 mg CQ following a presumptive initial treatment as recommended by the national malaria control programme (MOH). ANC services in health centres provide pregnant women with CQ and haematinics. The health centre 'Centre médical Paul VI' is a peri-urban health facility of Ouagadougou. It comprises general outpatient consultation service, paediatric and maternity wards, and a laboratory.Patients come from the peri-urban districts and the neighbouring villages.

Study design:

a) Comparative randomized trial.

Three groups will be studied. Pregnant women (primigravidae and secundigravidae from 12 to 24 weeks of pregnancy) will be randomly assigned, using random numbers lists, to treatment groups A to C as defined below:

* Group A : pregnant women receiving weekly 300 mg CQ prophylaxis after a curative dose (10mg/kg at days 1 and 2 +5mg/kg at day 3) at the first visit ;
* Group B : pregnant women receiving a presumptive CQ treatment at the 2nd and 3rd trimester of pregnancy (10mg/kg at days 1 and 2 +5mg/kg at day 3);
* Group C: pregnant women receiving a presumptive SP treatment at the 2nd and 3rd trimester of pregnancy (25mg sulfadoxine + 1,25mg pyrimethamine/kg in a single dose).

Another group composed of primiparous and secundiparous women who are not part of the study and who come to deliver at the health centre (group D) and who have not received chloroquine prophylaxis during pregnancy will be considered as reflecting the normal situation and act as a control group. These women will only be included during the first three months of the study.

At inclusion

1. personal information, anthropometric measures, clinical data, and obstetrical history, will be recorded
2. fingerprick blood will be collected for a thick and a thin blood smear, Hb and on filter paper for subsequent PCR tests
3. Treatment: The single dose of SP and the 3 days of CQ treatment will be administered supervised by the research team.

Study participants will be invited to come to the follow up visits or any time they feel sick or need health services.

Follow-up visits at the beginning of second and third trimester will include:

1. a clinical and parasitological examination. The health events since the previous visit will be recorded, Hb
2. providing chemoprophylaxis or treatment in accordance with the treatment group.

At delivery, the following data will be recorded:

1. delivery outcomes (birth weight, mode of delivery, APGAR score)
2. mother's peripheral blood for thick blood smear, Hb and filter paper for PCR
3. placental blood for thick blood smear, and collection on filter paper for PCR
4. cord blood for thick blood smear. If positive blood will be collected on filter paper for PCR

   b)Clinical trial for the assessment of clinical and parasitological efficacy of CQ and SP in pregnant women.

   Primigravidae and secundigravidae women presenting with an uncomplicated malaria attack will be randomly treated with CQ or SP and regularly followed up to assess clinical and parasitological efficacy. A molecular analysis of parasite gene mutations conferring resistance to chloroquine (PfCRT), and antifolates (DHFR, DHPS) will be performed.

   The patients will randomly assigned to treatment with either CQ or SP. They will then be followed-up during 28 days in accordance with WHO protocol. The follow up criteria are clinical (body temperature) and parasitological (peripheral parasitaemia).

   Sample size:

   a) Comparative randomized trial: Considering the prevalence of placenta parasitaemia to be 35% in pregnant women who do not get prophylaxis, 24% in women with weekly CQ prophylaxis, 15% in women with intermittent presumptive treatment with CQ and 5% in women with intermittent presumptive treatment with SP, and using a significance level of 5%, a power of 80% and 20% drop-out, each group should include 200 subjects.

   a) Drug efficacy assessment in pregnant women Considering the proportion of pregnant women with clinical failures to be 10-15% for chloroquine, and using a significance level of 5%, a power of 80% and 20% drop-out, a sample of 42 subjects should be included.

   Methods:
   1. Comparative randomized trial:

      Pregnant women will be recruited at the ANC unit of the health facility if fulfilling the following inclusion criteria and give oral informed consent.

      Inclusion criteria:
      * primi or secundigravidae - seen between 12th and 24th weeks of gestation
      * with a non 'at risk pregnancy' (multiple pregnancy, obstetric misproportions, previous caesarean, high blood pressure, diabetes, clinical signs of AIDS.
      * staying in a neighbouring district or village
      * ability to come for follow-up and delivery.

      Exclusion criteria:
      * At risk pregnancy
      * Severe systemic disease
      * Wish to withdraw from participation.

      Inclusion and follow-up procedures:

      The study aims and procedures will be clearly explained to those meeting the inclusion criteria.Enrolled women will be registered and a personal health file created, to be filled at enrolment, follow-up and, delivery. Each woman will be given a health record booklet to be presented at any visit. The following information will be recorded:

      At enrolment:
      * Identity number, date, and treatment group.
      * Name, age, profession, place of residence, address and name of husband and other close relatives.
      * Clinical history, axillary temperature, body weight, height, clinical anaemia, jaundice, splenomegaly, hepatomegaly, stethoscopy of heart and lungs, blood pressure and peripheral oedema)
      * Obstetrical data: date LMP, uterine size, presumed delivery date, foetal heart beat, previous pregnancy outcome (normal, abortion, stillbirth, complications during pregnancy and labour).
      * Biological data: Plasmodium species and density, Hb, filter paper blood for PCR.

      Follow-up:
      * Clinical follow-up: fever episodes, diseases, other treatments
      * Obstetrical follow-up: uterine height, foetal heart beat
      * Biological follow-up: Plasmodium species and density, Hb, filter paper blood for PCR.

      Delivery:

      - Date and time labor started, midwife's name.
      * Clinical data: body temperature, blood pressure, and clinical examination.
      * Mode of delivery, APGAR scores, and birthweight.
      * Biological data: mother's peripheral parasitaemia, haemoglobin concentration, placental parasitaemia, cord parasitaemia. Cord and mother's peripheral and placental blood collection on filter paper for PCR.

      Laboratory methods:

      - malaria diagnosis: a thick and thin smear of fingerprick blood will be prepared from each subject. Thin films will be fixed with methanol and stained with Giemsa in phosphate buffer (pH 7.2) for 30 min. and examined with a 100X oil immersion objective. The parasite species will be determined on the thin film and the parasites densities evaluated on the thick film by counting the number of asexual P.falciparum parasites against 200 leukocytes and expressed as number of parasites by microliter (µl) of blood assuming a standard leukocyte count of 8000/µl. At least 100 thick film fields will be examined to declare a slide negative.
      * Blood collection on filter paper: fingerprick blood will be collected on Whatmann 3MM chromatography filter paper. About 80-100 µl blood will be directly blotted on the paper strips, air dried and individually placed in plastic bag and conserved at room temperature in bottles containing silicagel.
      * HB will be measured using a HemoCue portable photometer.
      * Polymerase Chain Reaction (PCR) assays will be performed from blood on filter papers using the methods described by Jelinek et al., 1999, for resistance to antifolates and by Djimde et al.2001 for resistance to CQ.

      Drug efficacy assessment in pregnant women

      The subjects will be recruited at ANC and adult outpatient units of the health facility. Those who meet the inclusion criteria will be selected and requested to participate (oral informed consent) and then randomly allocated to CQ or SP treatment

      Inclusion criteria:

      • primi or secundigravidae from 12 to 24 weeks of gestation

      • pregnant women without 'at risk pregnancy'

      • axillary body temperature > 37.5°C and < 39.5°C

      • no clinical sign of severe malaria

      • mono infection of P. falciparum with a density > 2000 trophozoites /µl of blood
      * no sign of other febrile disease
      * staying in a neighbouring district or village

      Exclusion criteria:
      * severe malaria
      * any other febrile disease
      * previous side effects to CQ or SP consumption
      * loss to follow up.

      Inclusion and follow-up procedures:

      Enrolled women will be recorded with: date, identity number, name, age, profession, address, temperature, body weight, parasitaemia, haemoglobin concentration, treatment, follow-up temperatures, parasitaemia and Hb, other observations, and results of the test. Every subject will be asked to come at precise dates for follow up. Those lost of follow up will be actively searched for the next day.

      Methods:

      The WHO 28 days "assessment of therapeutic efficacy of antimalarials drugs for uncomplicated falciparum malaria in areas with intense transmission protocol" will be used, adapted to pregnant women.

      Data handling and statistical analysis All data will be recorded in pre-designed and tested questionnaires and/or registers. Then they will be progressively entered, cleared, checked and analysed using SPSS software.

      For the comparative randomized trial, a general analysis will aim to describe the study samples through the calculation of variables means (e.g. age, parity, parasite density, haemoglobin concentrations, birthweight), the frequency of some clinical data as malaria attacks, clinical results, delivery outcomes, mutations profiles.

      Then a comparative analysis will compare the proportions of main variables between the different treatment groups (peripheral, placenta, and cord blood parasitaemia, LBW, prevalence of resistant strains, mutations profiles, clinical and parasitological responses) using the chi-square test. The means (birthweight, haemoglobin concentrations, and number of clinical attacks) will be compared between groups by t-test and one way analysis of variance. Stratified or multivariate analysis tests will be used when necessary.

ELIGIBILITY:
Inclusion Criteria:

* primi or secundigravidae - seen between 12th and 24th weeks of gestation

  * with a non 'at risk pregnancy' (multiple pregnancy, obstetric misproportions, previous caesarean, high blood pressure, diabetes, clinical signs of AIDS.
  * staying in a neighbouring district or village
  * ability to come for follow-up and delivery.

Exclusion Criteria:

* • At risk pregnancy

  * Severe systemic disease
  * Wish to withdraw from participation.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 700
Dates: Start 2002-10; Primary Completion 2007-06 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
See detailed description

SECONDARY OUTCOMES:
see detailed description

CONTACTS AND LOCATIONS:
Overall Officials: Sheick O Coulibaly, MD, Principal Investigator — Laboratoire National de Sante Publique
Locations (1):
- Centre Medicale Paul VI, Ouagadougou, Ouagadougou, Burkina Faso

REFERENCES:
- See also: DBL-Centre for Health Resaerch and Development — http://www.dbl.life.ku.dk/